CLINICAL TRIAL: NCT00101166
Title: A Phase II Trial Using a Universal GM-CSF-Producing and CD40L-Expressing Bystander Cell Line (GM.CD40L) in the Formulation of Autologous Tumor Cell-Based Vaccines for Patients With Malignant Melanoma
Brief Title: Universal Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF)-Producing and CD40L Expressing Bystander Cell Line for Tumor Vaccine in Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Society of Clinical Oncology (Other); Society of Surgical Oncology (SSO) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13639; 0407-657 (Other: OBA)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2012-09

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — polyvalent melanoma cell vaccine; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine Therapy (Experimental): Treatment consisted of intradermal vaccine injections at 28-day intervals for a total of 3 immunizations. Injections were performed on Days 1, 29, and 57.
  Interventions: Biological: Bystander-Based Autologous Tumor Cell Vaccine

INTERVENTIONS:
Biological: Bystander-Based Autologous Tumor Cell Vaccine — The vaccine, consisting of one mL of cell suspension (GM.CD40L bystander cells admixed with an equivalent number of thawed autologous tumor cells), was administered into 8 separate injection sites, as described in treatment arm.
  Other Names: GM.CD40L; bystander cells; Melanoma Vaccine; Immunotherapy

SUMMARY:
The purpose of this study is to find out what effects (good and/or bad) this new cancer vaccine has on the patient and their cancer, whether it is safe and whether it can help get rid of their cancer (malignant melanoma). We want to check how the patient's immune system reacts, both before and after the vaccine treatment.

DETAILED DESCRIPTION:
The vaccine will be made by mixing two kinds of cells: 1) some of the patient's own malignant melanoma cells which were removed by surgery and then processed in the Cell Therapy Laboratory, and 2) experimental "bystander" cells. All the cells in the vaccine will be treated with high-dose X-rays to make sure that none of them grow and cause more cancer. The bystander cells, called "GM.CD40L", are human cells that have been genetically changed. The original cells, called K562, had the genes for human GM-CSF and CD40L inserted into them. These changes are designed to help boost the patient's immune system to better fight the cancer in their body.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIC or stage IV melanoma
* Measurable disease
* Age 18 or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* No radiation therapy within 2 weeks prior to first vaccine administration
* No chemotherapy within 4 weeks prior to first vaccine administration
* No steroid therapy within 4 weeks prior to first vaccine administration
* No surgery within 10 days prior to first vaccine administration
* Patient's written informed consent
* Patient's ability to comply with the visit schedule and assessments required by the protocol
* Adequate organ function (measured within a week of beginning treatment):

  * White blood count (WBC) > 3,000/mm^3 and absolute neutrophil count (ANC) >1500/mm^3
  * Platelets > 100,000/mm^3
  * Hematocrit > 25% and Hgb > 8 g/dL
  * Bilirubin < 2.0 mg/dL
  * Creatinine < 2.0 mg/dL, or creatinine clearance > 60 mL/min

Exclusion Criteria:

* Symptomatic or untreated brain metastasis
* Any serious ongoing infection
* Current corticosteroid or other immunosuppressive therapy
* Any other pre-existing immunodeficiency condition (including known HIV infection)
* Pregnant or lactating women -- Patients in reproductive age must agree to use contraceptive methods for the duration of the study (*A pregnancy test will be obtained before treatment)
* ECOG performance status of 2, 3, or 4
* Any second active primary cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Dessureault, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 patients with Stage IV melanoma were enrolled between November 2004 and May 2007. Fifteen of these patients did not receive any vaccine.
Groups:
- Vaccine Therapy: Treatment consisted of intradermal vaccine injections at 28-day intervals for a total of 3 immunizations. Injections were performed on Days 1, 29, and 57.
  Bystander-Based Autologous Tumor Cell Vaccine : The vaccine, consisting of one mL of cell suspension (GM.CD40L bystander cells admixed with an equivalent number of thawed autologous tumor cells), was administered into 8 separate injection sites, as described in treatment arm.
Period: Overall Study
Arm/Group | Vaccine Therapy
Started | 28
Completed | 18
Not Completed | 10
Not completed — progressive disease | 10

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 60 [24 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Related to Study Treatment
Description: Frequency of Study Related Toxicity. To evaluate the toxicity of the autologous tumor cell / GM.CD40L bystander cell vaccine. Toxicity was scored using the NCI Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE-3).
Time Frame: Average of 14 months
Population: All 28 participants who were vaccinated on this study.
Measure: Number; unit: participants
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 28
participants | 0

2. Primary Outcome: Number of Participants With Partial Response
Description: Response and progression were evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Average of 14 months
Population: All 28 participants who were vaccinated on this study.
Measure: Number; unit: participants
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 28
participants | 1

3. Secondary Outcome: Number of Participants With Stable Disease
Description: Patients with stable disease by RECIST criteria after 3 vaccine injections. Response and progression were evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Average of 14 months
Population: All 28 participants who were vaccinated on this study.
Measure: Number; unit: participants
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 28
participants | 8

4. Secondary Outcome: Time to Progression (TTP) in Months
Description: Response and progression were evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Progressive disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Average of 14 months
Population: All 28 participants who were vaccinated on this study.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 28
months | 3.8 [3 to 38]

5. Secondary Outcome: Overall Survival (OS) in Months
Description: Average overall survival time in months.
Time Frame: Average of 14 months
Population: All 28 participants who were vaccinated on this study.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 28
months | 12.8 [3 to 38]

ADVERSE EVENTS:
Time Frame: Average of 14 months. Every 4 weeks throughout the 4 month treatment phase and every 3 months thereafter.
Description: As in our Phase I study, there were no recorded systemic toxicities associated with the vaccine.
Arm/Group | Vaccine Therapy
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 10/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine Therapy (N=28)
Pain - Cardiac - Unrelated (Cardiac disorders) | 1 (1)
Transient localized erythema (Skin and subcutaneous tissue disorders) | 10 (10)
mild pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Localized depigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Induration (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the heterogeneity of the patient population, results were mainly descriptive in nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes